CLINICAL TRIAL: NCT03385590
Title: The Feasibility and Acceptability of a Soy-fiber-maize Blend Complementary Food and Its Effects on Stool Frequency, Stool Consistency, Microbiota Composition, Growth, and Dietary Intake of Children Aged 6 to 36 Months in Malawi.
Brief Title: Feasibility and Acceptability of a Soy-fiber-maize Complementary Food in Malawi.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB201700644
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Healthy
Keywords: healthy

STUDY DESIGN:
Intervention Model Description: Children 6-36 months will be fed soy-fiber-maize or soy-maize complementary foods for 6 months.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be blinded, on-site investigator will not be blinded due to the difficulty with blinding the foods. The off-site PI and outcome assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soy-fiber-maize (Experimental): Complementary food composed of soybean, soy fiber and maize flours.
  Interventions: Dietary Supplement: Soy-fiber-maize
- Maize (Active Comparator): Complementary food composed of maize flour.
  Interventions: Dietary Supplement: Maize

INTERVENTIONS:
Dietary Supplement: Soy-fiber-maize — Two servings of soy-maize porridge fortified with soy fiber (1.3 g per serving) will be consumed by the children each day for a period of six months.
  Arms: Soy-fiber-maize
Dietary Supplement: Maize — Two servings of maize porridge will be consumed by the children each day for a period of six months.
  Arms: Maize

SUMMARY:
The purpose of this intervention study is to assess the feasibility and acceptability of soy-fiber-maize versus soy-maize complementary foods on bowel movement frequency, transit time, growth, gastrointestinal symptoms, microbiota composition and activity.

DETAILED DESCRIPTION:
This is a 6-month randomized study to assess the feasibility and acceptability of soy-fiber-maize complementary food. Participants (caregiver/mother - child pairs) will complete a 2-week baseline period during which stool frequency, and stool consistency will be collected by paper questionnaire, and participants will collect a single stool. Dietary data will be obtained at baseline, 3 months and at 6 months during the study period. Participants will receive soy-fiber-maize or maize complementary foods twice a day for 6 months. Participants will attend a study visit every week for study food collection. During the study visit at baseline, 3 and 6 months, participants will complete a 24-hour dietary recall and height, weight and Mid Upper Arm Circumference will be measured on the children. At these same times, participants will provide stool samples. Participants will complete weekly questionnaires to assess gastrointestinal health, stool frequency and stool form. Furthermore, participants will participate in a focus group discussion at the end of the 6 months' study period to assess the feasibility and acceptability of soy-fiber-maize complementary foods for their children. Stool samples will be analyzed for differences in the microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Willing to have height and weight measured and provide demographic information (e.g age, race, sex).
* Willing to consume soy fiber or control porridge twice daily for a 6 months' period
* Willing to complete a weekly questionnaire throughout the entire 6 months' study.
* Willing to be interviewed for 24-Hour recall 3 times per 6 months' period throughout the study.
* Willing to provide 3 stool samples, one in each 2-weeks period throughout the study.

Exclusion Criteria:

* Have any known food allergies.
* Are currently taking medications for diarrhea.
* Have taken antibiotics within the past four weeks prior to randomization.
* Have more than 3 diarrheal episodes in the last week
* Currently participating in a clinical trial.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Compliance to feeding protocol | Weekly - baseline through 6 months
  Acceptability and feasibility of soy-fiber-maize blend versus maize only complementary food as measured by compliance to feeding complementary food.

SECONDARY OUTCOMES:
Stool consistency | Weekly - baseline through 6 months
  Stool consistency rating by Modified Bristol Stool Form Scale for Children, scale of 1-5, = with fewer 4 and 5 scores considered improvment.
Number of bowel movements | Weekly - baseline through 6 months
  Number of bowel movements per week
Microbiota profile changes | Baseline, month 3 and month 6
  Percent change at phylum and genus levels; changes in OTUs
Growth | Baseline, month 3 and month 6
  Increase in height, weight and Mid Upper Arm Circumference
Dietary intake | Baseline, month 3 and month 6
  24-hour dietary recall assessing intake of children

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Dahl, PhD, Principal Investigator — University of Florida
Locations (1):
- Kabudula Community Hospital, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Undecided